CLINICAL TRIAL: NCT03108092
Title: Health Economic Evaluation Alongside the OPERAM Trial (OPtimising thERapy to Prevent Avoidable Hospital Admissions in the Multimorbid Older People: a Cluster Randomised Controlled Trial).
Brief Title: Health Economic Evaluation Alongside the OPERAM Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Cork University Hospital (Other); UMC Utrecht (Other); University of Basel (Other); Université Catholique de Louvain (Other); Utrecht University (Other); University of Bern (Other); State Secretariat for Education Research and Innovation, Switzerland (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-01200_1
Record Dates: First submitted 2017-04-04; First posted 2017-04-11 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: 3 or More Chronic Conditions for 6 Months or Longer; 5 or More Regular Drugs
Keywords: Drug Utilization Review; Older people; Health economics
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRIP intervention (Experimental): The intervention will take place during the initial hospital admission (Index Hospitalisation) or an equivalent situation for outpatients. STRIP is a structured method to perform pharmacotherapy optimisation. The STRIP-intervention consists of 9 steps.
  Interventions: Other: STRIP intervention
- Control (Sham Comparator): Participants in the control group will receive medication review by the prescribing physicians in accordance with usual care. If an extended drug review is in place in a ward/specialty corresponding characteristics are collected on cluster level.
  Interventions: Other: Control

INTERVENTIONS:
Other: STRIP intervention — The STRIP intervention consists of 9 steps: 1. structured history taking of medication 2. recording medication and diagnoses in STRIPA 3. structured drug review based on the STRIPA with the integrated Screening Tool of Older Person's Prescriptions (STOPP)/ Screening Tool to Alert Doctors to the Right Treatment (START) criteria 4. communication and discussion of the structured drug review with prescribing physician with possible adaptation of the recommendation 5. shared decision-making with the patient with possible adaptation of the recommendation 6. optional revision based on new accumulating data during hospitalisation (e.g. new diagnoses, adverse drug reactions) 7. generation of general practioner (GP) report 8. delivery of the report to the patient and to the GP (optional additional direct communication) 9. follow-up
  Other Names: Systematic drug review
  Arms: STRIP intervention
Other: Control — Standard care in the department where the trial is conducted
  Other Names: Standard care
  Arms: Control

SUMMARY:
The objective of the health economic evaluation is to perform a state-of-the-art economic analysis of the STRIP intervention, alongside the OPERAM Randomised Controlled Trial (RCT).

DETAILED DESCRIPTION:
Background:

Drug-related morbidity and mortality is an increasing problem in European healthcare systems. Multimorbidity, polypharmacy and old age are important risk factors for drug-related hospital admissions (DRAs). The reported incidence of DRAs in the elderly may be as high as 30% of all acute cases, and about half of DRAs are likely to be preventable. They are mainly related to prescribing problems and non-compliance with drug regimens, and are very costly. Public funds spent on prescription medicines are steadily increasing in many European countries. Under strained budget conditions, healthcare services need to show that they provide value for money, and thus detailed health economic evaluations have become essential for health budget planning. Some studies assessing the impact of medication optimising interventions have assessed the cost-effectiveness of such interventions. A recent Cochrane review looking at interventions to optimise prescribing for the older people in care homes found an unclear effect of interventions on drug costs (Alldred DP 2013). Further assessment of healthcare costs related to inappropriate medication and the cost-effectiveness of pharmacotherapy optimising solutions is essential for a better control of rapidly increasing health care costs.

Design:

European multi-centre, cluster randomised, controlled trial of people aged 70 years or older, with multimorbidity and polypharmacy, being on an ambulatory visit or on a hospital stay in one of the four participating centres in Ireland, Belgium, Switzerland and the Netherlands. A cluster is defined around a treating physician, i.e. the treating physician is randomised and defines the allocation of his patients. Clusters of patients will be randomised to the intervention arm receiving STRIP for optimising therapy or to the control arm undergoing usual clinical care. The patients of physicians who are allocated to the intervention group will undergo a systematic drug review and pharmacotherapy optimisation by a physician and a pharmacist using STRIP, including the STRIPA software. That provides the research team with a recommendation of changes in the patient's medication. Based on STRIPA recommendation and agreement on changes to the patients' pharmacotherapy between the team of the research physician and pharmacist and the prescribing physician, will the patient receive structured counselling about his/her medication; general practitioners will receive a report. Health economic data (covering medical resource use, the provision of informal care and health-related quality of life using the EQ-5D instrument) will be collected from enrolled patients at baseline and during the follow-up phone calls after 2, 6 and 12 months. Patients will be asked to complete a booklet serving as a memory aid. Where relevant, information can also be provided by proxy respondents (e.g. family members, primary care physicians). Additionally, staff time spent on the intervention and comparable activities in the comparator arm will be collected from site staff.

Objectives:

The objectives of the health-economic evaluation are to assess the impact of pharmacotherapy optimisation by the STRIP intervention on economic parameters, health care utilisation and preference-based quality of life.

Statistical considerations:

Over all sites, 80 clusters with a cluster size ranging from 12 to 38 participants will be included. Therefore, 2000 patients, 1000 patients in each arm, will be recruited over 18 months. Health economic analyses will comprise the assessment of cost differences between the trial arms, of differences in quality-adjusted lifetime between the trial arms (expressed as quality-adjusted life years), and of the incremental cost-effectiveness of the intervention in comparison with the comparator, i.e. standard care.

Cost will be calculated by combining the healthcare resource utilisation observed in the trial with national unit costs from sources external to the trial. Health economic analyses involving costs are necessarily country-specific. It is planned to perform these analyses for at least two countries contributing patients to the OPERAM trial, which remain to be specified. This will involve the use of all or a subset of trial data (depending on the degree of heterogeneity observed between participating countries) in combination with a set of national unit costs and a national valuation algorithm for the EQ-5D. Perspectives of cost assessment remain to be decided. Typical perspectives are those of the healthcare system or a nationally relevant third party payer.

All health economic analyses will be subjected to extensive sensitivity analyses to understand the robustness of the results given stochastic uncertainty inherent in the trial data and parameter uncertainty expected for the external unit cost data.

Additionally, performance characteristics of the 5-level version (used in all patients) and the 3-level version (additionally administered in a subsample of 300 patients of the EQ-5D will be compared, e.g. in terms of discriminatory power, responsiveness to change over time and effect size.

ELIGIBILITY:
Inclusion Criteria:

* People 70 years of age or older
* Multimorbidity: 3 or more coexistent chronic conditions defined by 3 distinct International Classification of Diseases (ICD-10) codes with an estimated duration of 6 months or more or based on a clinical decision
* Polypharmacy i.e. five or more different regular drugs (defined as authorised medications with registration numbers) for more than 30 days.
* Estimated minimal length of stay within the cluster is sufficient to apply the intervention
* If outpatient: prescribing physician has GP function and has a planned appointment to conduct intervention

Exclusion Criteria:

* Inability to provide informed consent or to obtain informed consent from a proxy for patients with cognitive impairment
* Direct admission to palliative care (< 24h after admission)
* Has passed or will pass a systematic structured drug review during this hospitalisation or within the last two months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2009 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The cost-effectiveness of the STRIP intervention | 12 months
  The cost-effectiveness analysis (CEA) is performed by combining clinical data, quality of life data and healthcare utilisation data collected within the trial, and unit costs for participating countries that will stem from external sources.

SECONDARY OUTCOMES:
Healthcare utilisation | 12 months
Informal care received | 12 months
Healthcare costs | 12 months
  Performed during the follow-up period, based on unit costs for participating countries that will stem from external sources
Quality of life EQ-5D | 2, 6, and 12 months
  Measured by the 5-level version of the European Quality of Life-5 Dimensions questionnaire (EQ-5D)
Direct costs of the STRIP intervention | during the index hospitalisation at baseline

OTHER OUTCOMES:
Exploratory outcome measures | 12 months
  Extrapolation of CEA beyond 12 months may be performed to cover longer-term effects of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, Prof., Study Chair — Head of Ambulatory Care Department of General Internal Medicine Inselspital, Bern University Hospital, University of Bern, Switzerland
Locations (4):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Dept. of Medicine (Geriatrics), University College Cork, Cork, Ireland
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- University of Bern and University Hospital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laws MB. Adverse drug reactions as cause of admission to hospital: definition of adverse drug reactions needs to include overdose. BMJ. 2004 Aug 21;329(7463):459-60; author reply 460. doi: 10.1136/bmj.329.7463.459-b. No abstract available. PMID 15321917
- [Result] Leendertse AJ, Egberts AC, Stoker LJ, van den Bemt PM; HARM Study Group. Frequency of and risk factors for preventable medication-related hospital admissions in the Netherlands. Arch Intern Med. 2008 Sep 22;168(17):1890-6. doi: 10.1001/archinternmed.2008.3. PMID 18809816
- [Result] Gillespie U, Alassaad A, Henrohn D, Garmo H, Hammarlund-Udenaes M, Toss H, Kettis-Lindblad A, Melhus H, Morlin C. A comprehensive pharmacist intervention to reduce morbidity in patients 80 years or older: a randomized controlled trial. Arch Intern Med. 2009 May 11;169(9):894-900. doi: 10.1001/archinternmed.2009.71. PMID 19433702
- [Result] Howard RL, Avery AJ, Slavenburg S, Royal S, Pipe G, Lucassen P, Pirmohamed M. Which drugs cause preventable admissions to hospital? A systematic review. Br J Clin Pharmacol. 2007 Feb;63(2):136-47. doi: 10.1111/j.1365-2125.2006.02698.x. Epub 2006 Jun 26. PMID 16803468
- [Result] Alldred DP, Raynor DK, Hughes C, Barber N, Chen TF, Spoor P. Interventions to optimise prescribing for older people in care homes. Cochrane Database Syst Rev. 2013 Feb 28;(2):CD009095. doi: 10.1002/14651858.CD009095.pub2. PMID 23450597